CLINICAL TRIAL: NCT00934570
Title: Reduction of Adolescent Risk Factors for Type 2 Diabetes and Cardiovascular Disease
Brief Title: Activity and Metformin Intervention in Obese Adolescents
Acronym: REACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Cheryl, Dr Cheril Clarson, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-08-259; 15590 (Other: REB)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Metformin; Physical activity; Cardiovascular health
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Motor Activity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metformin, Standard exercise (Active Comparator): Lifestyle intervention with metformin and standard exercise program.
  Interventions: Drug: Metformin and standard exercise
- Placebo, Standard exercise (Placebo Comparator): Lifestyle intervention with placebo and standard exercise program
  Interventions: Behavioral: Placebo Standard exercise
- Metformin, Intensive exercise (Active Comparator): Lifestyle intervention with metformin and intensive exercise
  Interventions: Drug: Metformin Intensive exercise
- Placebo, Intensive exercise (Placebo Comparator): Lifestyle intervention with placebo and intensive exercise program.
  Interventions: Behavioral: Intensive exercise

INTERVENTIONS:
Drug: Metformin and standard exercise — Metformin 1500 mg daily for 2 years
  Other Names: GlumetzaTM 500 mg Extended Release
  Arms: Metformin, Standard exercise
Drug: Metformin Intensive exercise — Metformin 1500 mg daily for 2 years
  Other Names: GlumetzaTM 500 mg Extended Release
  Arms: Metformin, Intensive exercise
Behavioral: Placebo Standard exercise — Standard exercise
  Arms: Placebo, Standard exercise
Behavioral: Intensive exercise — Placebo Intensive exercise
  Arms: Placebo, Intensive exercise

SUMMARY:
The purpose of this study is to assess the sustainability of a two-year intervention aimed at improving body mass index (BMI) and metabolic and vascular health in obese youth. The study will compare lifestyle changes with diet and exercise alone with changes in lifestyle in combination with metformin medication. An initial intensive exercise program will also be compared with a standard exercise program.

Hypothesis: Metformin therapy in combination with intensive lifestyle intervention in obese children and adolescents will be associated with reduced rate of weight gain, improved BMI, body composition, physical activity, physical fitness, insulin sensitivity, blood lipid profiles, adipocytokines and vascular function.

DETAILED DESCRIPTION:
This study will assess the sustainability of a two-year intervention and the degree of improvement in body mass index (BMI) and reduction in risk factors for type 2 diabetes and diabetes related cardiovascular disease, as well as evaluating the additive effect of metformin (as GlumetzaTM 500 mg Extended Release Tablets) and comparing an initial intensive exercise program with a standard exercise program. The study will recruit obese youth who are at risk for type 2 diabetes and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescents defined as BMI greater than the 95th percentile for age and gender
* Metformin naive subjects

Exclusion Criteria:

* Elevated fasting plasma glucose ≥ 6.0 mmol/L
* 2 hour plasma glucose ≥ 11.1 mmol/L after a standard glucose load
* A1C > 6.0%
* Medication other than "over the counter" drugs, oral contraceptive pill or thyroid hormone replacement
* Smoking
* Pregnancy
* Renal insufficiency (serum creatinine > the upper limit of normal)
* Hepatic dysfunction (> 1.5 times the upper limit of normal for AST and ALT)
* Latex Allergy
* Hypersensitivity to metformin or its ingredients
* Breast feeding
* Subjects with a history of lactic acidosis
* Abnormal creatinine clearance
* HIV, HBV, and HCV infections
* Drug and alcohol abuse
* Severe mental disorders
* Subjects who are planning radiologic exams involving in i.v. injection of iodinated contract materials
* Participation in another clinical trial
* Significant history or presence of cardiovascular, pulmonary, gastrointestinal, immunologic, endocrine, neurologic disorders
* Malignant diseases
* Previous exposure to any pharmaceutical antidiabetic agent

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Reduction in BMI | 2 years

SECONDARY OUTCOMES:
Improvement in physical activity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheril Clarson, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Clarson CL, Brown HK, De Jesus S, Jackman M, Mahmud FH, Prapavessis H, Robinson T, Shoemaker JK, Watson M, Dowd AJ, Hill DJ. Effects of a Comprehensive, Intensive Lifestyle Intervention Combined with Metformin Extended Release in Obese Adolescents. Int Sch Res Notices. 2014 Nov 10;2014:659410. doi: 10.1155/2014/659410. eCollection 2014. PMID 27433488
- [Derived] Wilson AJ, Prapavessis H, Jung ME, Cramp AG, Vascotto J, Lenhardt L, Shoemaker JK, Watson M, Robinson T, Clarson CL. Lifestyle modification and metformin as long-term treatment options for obese adolescents: study protocol. BMC Public Health. 2009 Nov 30;9:434. doi: 10.1186/1471-2458-9-434. PMID 19943971
- See also: Click here for more information about this study: Metformin and Activity Intervention in Obese Adolescents — http://www.lhsc.on.ca/About_Us/LHSC/News_Events/Healthy_Eating_and_Activity.htm